CLINICAL TRIAL: NCT02700360
Title: A Randomized, Open-Label, Single -Dose, Crossover, Phase I Clinical Trial to Evaluate the Effect of Food on the Safety, Tolerability and Pharmacokinetics of EC-18 After Oral Administration in Healthy Volunteers
Brief Title: Evaluation of the Food Effect on the Safety, Tolerability, PK of EC-18 After Oral Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enzychem Lifesciences Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: EC18-102
Record Dates: First submitted 2016-01-20; First posted 2016-03-07 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-03

CONDITIONS: Chemotherapy-Induced Neutropenia
Keywords: EC-18; Hematology; Cancer; Neutropenia
MeSH Terms: conditions — Neoplasms; Neutropenia | interventions — Diet, High-Fat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part 1(1,000mg dose): group 1 (Experimental): period 1: EC-18 1,000 mg(500 mg/cap, 2 capsules) once daily, after high-fat diet intake; period 2: EC-18 1,000 mg(500 mg/cap, 2 capsules) once daily, on an empty stomach; cross-over period: 7 days
  Interventions: Dietary Supplement: high-fat diet; Drug: EC-18
- Part 1(1,000mg dose): group 2 (Experimental): period 1: EC-18 1,000 mg(500 mg/cap, 2 capsules) once daily, on an empty stomach; period 2: EC-18 1,000 mg(500 mg/cap, 2 capsules) once daily, after high-fat diet intake; cross-over period: 7 days
  Interventions: Dietary Supplement: high-fat diet; Drug: EC-18
- Part 2(500mg dose): group 3 (Experimental): period 1: EC-18 500 mg(500 mg/cap, 1 capsule) once daily, after high-fat diet intake; period 2: EC-18 500 mg(500 mg/cap, 1 capsule) once daily, on an empty stomach; cross-over period: 7 days
  Interventions: Dietary Supplement: high-fat diet; Drug: EC-18
- Part 2(500mg dose): group 4 (Experimental): period 1: EC-18 500 mg(500 mg/cap, 1 capsule) once daily, on an empty stomach; period 2: EC-18 500 mg(500 mg/cap, 1 capsule) once daily, after high-fat diet intake; cross-over period: 7 days
  Interventions: Dietary Supplement: high-fat diet; Drug: EC-18
- Part 2(2,000mg dose): group 5 (Experimental): period 1: EC-18 2,000 mg(500 mg/cap, 4 capsules) once daily, after high-fat diet intake; period 2: EC-18 2,000 mg(500 mg/cap, 4 capsules) once daily, on an empty stomach; cross-over period: 7 days
  Interventions: Dietary Supplement: high-fat diet; Drug: EC-18
- Part 2(2,000mg dose): group 6 (Experimental): period 1: EC-18 2,000 mg(500 mg/cap, 4 capsules) once daily, on an empty stomach; period 2: EC-18 2,000 mg(500 mg/cap, 4 capsule) once daily, after high-fat diet intake; cross-over period: 7 days
  Interventions: Dietary Supplement: high-fat diet; Drug: EC-18

INTERVENTIONS:
Dietary Supplement: high-fat diet — This trial is conducted as a randomized, open-label, single -dose, crossover, phase I to evaluate the effect of food on the safety, tolerability and pharmacokinetics of EC-18. EC-18 is given at an oral, once daily in condition of empty stomach and a high fat diet(900~1,000 kcal, contains 50~60%lipid).This trial is divided into Part 1(1,000mg dose) and Part 2(500mg dose and 2,000mg dose), 12 subjects are included in each dose and cross-over period is 7 days. After Part 1 study, If primary PK parameters of EC-18 is affected by food and AEs meeting study discontinuation criteria are not reported, Part 2 will proceed in consecutive order with registering new subjects.
Drug: EC-18 — This trial is conducted as a randomized, open-label, single -dose, crossover, phase I to evaluate the effect of food on the safety, tolerability and pharmacokinetics of EC-18. EC-18 is given at an oral, once daily in condition of empty stomach and a high fat diet(900~1,000 kcal, contains 50~60%lipid).This trial is divided into Part 1(1,000mg dose) and Part 2(500mg dose and 2,000mg dose), 12 subjects are included in each dose and cross-over period is 7 days. After Part 1 study, If primary PK parameters of EC-18 is affected by food and AEs meeting study discontinuation criteria are not reported, Part 2 will proceed in consecutive order with registering new subjects
  Other Names: EC18 Soft-capsule

SUMMARY:
A Randomized, Open-Label, Single -Dose, Crossover, Phase I Clinical Trial to Evaluate the Effect of Food on the Safety, Tolerability and Pharmacokinetics of EC-18 after Oral Administration in Healthy Volunteers

DETAILED DESCRIPTION:
In vitro and in vivo efficacy studies and clinical trials have shown that EC-18 has a mode of action of improving neutropenia by promoting neutrophil production from hematopoietic stem cells and at the same time, efficiently controlling STAT6/Complement 3(C 3), suggesting its potential to be developed as an orally administered new drug for treatment of neutropenia resulting from decreased neutrophils caused by administration of an anticancer agent.

This study is a randomized, open-Label, single -dose, crossover, phase I clinical trial to evaluate the effect of food on the safety, tolerability and pharmacokinetics of EC-18 after oral administration in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult aged between 19 and 45 years, inclusive, at the time of providing the informed consent form
2. body weight: ≥ 55kg(male), ≥ 50kg(female)
3. BMI: 18.5 kg/m2 ≦ BMI < 25.0 kg/m2 [BMI(body mass index) = Body weight (kg)/[height (m)]2 ]
4. in female subjects, the result of serum β-hCG pregnancy test comes out negative at screening, urine β-hCG test comes out negative before taking medication during the period set by this protocol have to be included one of the below conditions.

   * postmenopausal(no natural menstruation at least 2 years)
   * surgically sterile(hysterectomy or bilateral ovariotomy, tubal ligation or sterile condition by other ways)
   * sterility of male partner before screening(proof the azoospermia after vasectomy), and this is the only partner of the subject.
   * agree with using a proper and continuous method of contraception start on 14 days(at least) before the1st IND administration and for 28 days(at least) after the last IND administration

     * proper contraception means physical barrier method including condom, contraceptive diaphragm or cervix cap, do not use a hormones including contraceptive or oral contraceptive during the study.
5. if the male have a sex life with childbearing aged female, maintain proper contraception during the study and for 28 days after the last IND administration, agree with "do not donate the sperm"(if the female partner is infertility, above contraceptions are not necessary)
6. Written consent on voluntary decision of participation and compliance with precautions after being fully informed of and completely understanding this trial

Exclusion Criteria:

1. Hypersensitivity to a drug containing an ingredient of the investigational product(EC-18) or similar ingredient (e.g., deer antler) or other drugs (e.g., aspirin, antibiotics) or medical history of clinically significant hypersensitivity
2. Active infection such as chronic or local infection based on screening tests or inquiry, verifiable medical records
3. Serious infection that required hospitalization or use of antibiotics within 30 days prior to the first dose of the investigational product, based on an inquiry or verifiable medical records
4. Presence of a clinically significant hepatic, renal, gastrointestinal, respiratory, musculoskeletal, endocrine, nervous, blood, cardiovascular, urogenital, psychiatric disorder or its prior history
5. (1) Presenting tuberculosis or prior history of tuberculosis or (2) positive results from a QuantiFERON®-TB Gold in Tube Assay conducted due to a contact with a tuberculosis patient within the past 3 months or signs and symptoms of suspected tuberculosis
6. Prior history of a gastrointestinal disorder (e.g., Crohn's disease, ulcer) or surgery (except for simple appendectomy or hernia surgery) that may affect drug absorption, etc.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
evaluate safety and tolerability: Number and severity of ADRs monitoring such as subjective, objective symptom(change value from baseline) | Day-3(Day5), Day-2(Day6), Day-1(Day7), Day1(Day8), Day2(Day9), D3(Day10) and Day15(follow-up)
evaluate safety and tolerability:vital sign(change value from baseline) | screening, 0(before medication) of Day-3(Day5), Day-2(Day6), Day-1(Day7), Day1(Day8), after medication 4, 12, 24, 36, 48hours and Day15(Follow-up)
evaluate safety and tolerability: physical examination(change value from baseline) | screening, Day-3(Day5), Day3(Day10) and Day15(follow-up)
evaluate safety and tolerability: clinical laboratory test(change value from baseline) | screening, Day-3(Day5), Day3(Day10) and Day15(follow-up)
evaluate safety and tolerability: EKG(change value from baseline) | screening, Day-3(Day5) and Day15(follow-up)

SECONDARY OUTCOMES:
evaluate pharmacokinetics: Cmax | 33 times per each period, total 66 times; Day-2(Day6):0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48hours; Day1(Day8):0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48hours
evaluate pharmacokinetics: AUClas | 33 times per each period, total 66 times; Day-2(Day6):0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48hours; Day1(Day8):0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48hours
evaluate pharmacokinetics: tmax | 33 times per each period, total 66 times; Day-2(Day6):0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48hours; Day1(Day8):0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48hours
evaluate pharmacokinetics: AUCinf | 33 times per each period, total 66 times; Day-2(Day6):0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48hours; Day1(Day8):0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48hours
evaluate pharmacokinetics: t1/2 | 33 times per each period, total 66 times; Day-2(Day6):0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48hours; Day1(Day8):0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48hours
evaluate pharmacokinetics: CL/F | 33 times per each period, total 66 times; Day-2(Day6):0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48hours; Day1(Day8):0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48hours
evaluate pharmacokinetics: Vd/F | 33 times per each period, total 66 times; Day-2(Day6):0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48hours; Day1(Day8):0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 14, 16, 24, 36, 48hours

CONTACTS AND LOCATIONS:
Overall Officials: Min-Soo Park, Professor, Principal Investigator — Yonsei University Health System, Severance Hospital (Seoul)
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No